CLINICAL TRIAL: NCT06773351
Title: A Response Surface Analysis for the Interaction Between Ciprofol and Sevoflurane During Anesthesia Induction
Brief Title: A Response Surface Analysis for the Interaction Between Ciprofol and Sevoflurane
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Feng Gao (Other)
Collaborators: Sichuan Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ-IRB202412125; S219 (Other Grant/Funding Number: Beijing Kangmeng Charity Foundation)
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Induction of General Anesthesia
Keywords: ciprofol; response surface analysis
MeSH Terms: interventions — Sevoflurane; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sevoflurane group (Experimental): Sevoflurane doses were 0,0.7, 1.0, 1.5, 2.0, 2.5%
  Interventions: Drug: Sevoflurane 0 + different doses of ciprofol; Drug: Sevoflurane 0.7% + different doses of ciprofol; Drug: Sevoflurane 1.0% + different doses of ciprofol 0.05; Drug: Sevoflurane 1.5% + differnet doses of ciprofol; Drug: Sevoflurane 2.0% + different doses of ciprofol; Drug: Sevoflurane 2.5% + different doses of ciprofol
- ciprofol group (Experimental): The doses of ciprofol were 0, 0.05, 0.1, 0.2, 0.3, 0.4mg/kg
  Interventions: Drug: Ciprofol 0 + different end-expiratory concentration of sevoflurane; Drug: Ciprofol 0.05mg/kg + different end-expiratory concentration of sevoflurane; Drug: Ciprofol 0.1mg/kg + different end-expiratory concentration of sevoflurane; Drug: Ciprofol 0.2 mg/kg + different end-expiratory concentration of sevoflurane; Drug: Ciprofol 0.3 mg/kg + different end-expiratory concentration of sevoflurane; Drug: Ciprofol 0.4 mg/kg + different end-expiratory concentration of sevoflurane

INTERVENTIONS:
Drug: Sevoflurane 0 + different doses of ciprofol — Sevoflurane 0% combined with ciprofol 0.1, 0.2, 0.3, 0.4, 0.6mg/kg, respectively.
  Arms: sevoflurane group
Drug: Sevoflurane 0.7% + different doses of ciprofol — Sevoflurane 0.7% combined with ciprofol 0.1, 0.2, 0.3, 0.4, 0.5mg/kg, respectively.
  Arms: sevoflurane group
Drug: Sevoflurane 1.0% + different doses of ciprofol 0.05 — Sevoflurane 1.0% combined with ciprofol 0.05, 0.1, 0.2, 0.3, 0.4mg/kg, respectively.
  Arms: sevoflurane group
Drug: Sevoflurane 1.5% + differnet doses of ciprofol — Sevoflurane 1.5% combined with ciprofol 0.05, 0.1, 0.2, 0.3, 0.4mg/kg, respectively.
  Arms: sevoflurane group
Drug: Sevoflurane 2.0% + different doses of ciprofol — Sevoflurane 2.0% combined with ciprofol 0.05, 0.1, 0.15, 0.2, 0.3mg/kg, respectively.
  Arms: sevoflurane group
Drug: Sevoflurane 2.5% + different doses of ciprofol — Sevoflurane 2.5% combined with ciprofol 0.05, 0.1, 0.15, 0.2, 0.3mg/kg, respectively.
  Arms: sevoflurane group
Drug: Ciprofol 0 + different end-expiratory concentration of sevoflurane — Ciprofol 0 combined with sevoflurane 0.7, 1.5, 2.0, 2.5, 3.5%, respectively.
  Arms: ciprofol group
Drug: Ciprofol 0.05mg/kg + different end-expiratory concentration of sevoflurane — Ciprofol 0.05 mg/kg combined with sevoflurane 0.7, 1.5, 2.0, 2.5, 3.5 %, respectively.
  Arms: ciprofol group
Drug: Ciprofol 0.1mg/kg + different end-expiratory concentration of sevoflurane — Ciprofol 0.1mg/kg combined with sevoflurane 0.5, 1.5, 2.0, 2.5, 3.0 %, respectively.
  Arms: ciprofol group
Drug: Ciprofol 0.2 mg/kg + different end-expiratory concentration of sevoflurane — Ciprofol 0.2 mg/kg combined with sevoflurane 0.5, 1.5, 2.0, 2.5, 3.0 %, respectively.
  Arms: ciprofol group
Drug: Ciprofol 0.3 mg/kg + different end-expiratory concentration of sevoflurane — Ciprofol 0.3 mg/kg combined with sevoflurane 0.5, 1.0, 1.5, 2.0, 2.5 %, respectively.
  Arms: ciprofol group
Drug: Ciprofol 0.4 mg/kg + different end-expiratory concentration of sevoflurane — Ciprofol 0.4 mg/kg combined with sevoflurane 0.5, 1.0, 1.5, 2.0, 2.5 %, respectively.
  Arms: ciprofol group

SUMMARY:
Intravenous and inhalation combined anesthesia is a commonly used method for maintaining general anesthesia in clinical practice. This study aims to explore the interaction between ciprofol and sevoflurane. By employing response surface methodology, we constructed a three-dimensional pharmacodynamic interaction surface for various dose combinations of ciprofol and sevoflurane. This approach allows us to determine the nature of the interaction between the two drugs at any given level, thereby providing a ciprofol understanding of the dose-response relationship when ciprofol and sevoflurane are used in combination. This knowledge will serve as a theoretical basis for rational drug administration during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective general anesthesia and non-cardiac surgery;
* Age 18-60 years old, gender is not limited;
* ASA I or II level;
* Body mass index (BMI) 18-30 kg/m2

Exclusion Criteria:

* Preoperative assessment of potential difficult airway risk;
* Airway hyperreactivity;
* There is disease of the central nervous system or cardiovascular system;
* Currently using drugs that may alter the pharmacokinetics and pharmacokinetics of the drug under study;
* Known or suspected allergy or contraindication to the components or regimens of the investigational drug;
* A history of drug or alcohol addiction;
* Patients with gastroesophageal reflux disease;
* Severe liver and kidney dysfunction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bispectral Index (BIS) value | Induction period of anesthesia
  The BIS usually ranges from 0 to 100, with 0-20 indicating a state of deep anesthesia or coma; 20-40 indicates moderate anesthesia; 40-60 indicates mild anesthesia; 60-80 indicates sedation; 80-100 indicates wakefulness.
The score of Observer's Assessment of Alertness/Sedation Scale | Induction period of anesthesia
  The Observer's Assessment of Alertness/Sedation (OAAS) scale ranges from 1 to 5 points.
  5 (awake) : The patient responds quickly to the name call with normal intonation, normal verbal answers, normal facial expressions, and bright eyes without drooping.
  4 (mild sedation) : The patient is slow to respond to the name call in normal intonation, the verbal answer is slightly slow or vague, the facial expression is slightly relaxed, the eyes are glassy and the upper eyelid is slightly droopy.
  3 (moderate sedation) : The patient responds only to the name call out loud, verbal responses are significantly slower or slower, facial expressions are significantly relaxed, and eyes are fixed with a visibly droopy upper eyelid.
  2 (deep sedation) : The patient responds only to nudging or shaking, and the verbal response is indistinct.
  1 (deep sleep, unconscious) : The patient does not respond to nudging or shaking.
  An OAA/S score of 2-5 is considered a response.
Numbers of of participants with laryngoscopy and tracheal intubation positive response | Induction period of anesthesia
  Laryngoscopic exposure of the glottis to obtain Cormack-Lehane level 1 or 2 visual field and maintain it for 5 seconds: verbal response, eye opening, painful expression, coughing, retraction, or other purposeful or unpurposeful movements are considered responsive.
Numbers of participants with tracheal intubation stress positive respose | Induction period of anesthesia
  If the increase in heart rate (HR) or mean arterial pressure (MAP) compared to the baseline value was greater than or equal to 15% during this procedure, the stress response induced by tracheal intubation was considered to have failed to be effectively suppressed, and the effect was recorded as 1.
Blood plasma concentration | Induction period of anesthesia

SECONDARY OUTCOMES:
HR | Period of anesthesia
  For adults, the normal heart rate range is usually between 60 and 100 beats per minute. During anesthesia, HR less than 20% of baseline is considered hypotensive
MAP | Period of anesthesia
  The normal range of MAP is usually 70-105 mmHg. MAP is one of the important indicators to measure the function of the human circulatory system, which represents the average arterial blood pressure in a cardiac cycle. During anesthesia, MSP less than 20% of baseline is considered hypotensive.
Adverse reactions | Perioperative period